CLINICAL TRIAL: NCT02119663
Title: A Randomized, Double-Blind, Phase 3 Study of the JAK 1/2 Inhibitor Ruxolitinib or Placebo in Combination With Capecitabine in Subjects With Advanced or Metastatic Adenocarcinoma of the Pancreas Who Have Failed or Are Intolerant to First-Line Chemotherapy (The JANUS 2 Study)
Brief Title: A Study of Ruxolitinib in Pancreatic Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The safety committee found no safety issues but recommended halting the study based on a lack of efficacy in a similar trial. The sponsor terminated the trial.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-363
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ruxolitinib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib plus capecitabine (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Capecitabine
- Placebo plus capecitabine (Active Comparator)
  Interventions: Drug: Placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets to be administered by mouth twice daily (BID)
  Other Names: Jakafi ®; Jakavi ®
  Arms: Ruxolitinib plus capecitabine
Drug: Placebo — 5 mg matching placebo tablets to be administered by mouth twice daily (BID)
  Arms: Placebo plus capecitabine
Drug: Capecitabine — 150 mg or 500 mg tablets to be administered by mouth twice daily (BID)

SUMMARY:
This was to determine the efficacy, based upon overall survival, of ruxolitinib added to capecitabine for the treatment of metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This was a randomized, double-blinded, placebo-controlled, Phase 3 study, in which approximately 270 participants with advanced or metastatic adenocarcinoma of the pancreas who had failed or were intolerant to first-line chemotherapy were to be randomized (1:1) to one of the following treatment groups:

* Treatment A (N = 135): Capecitabine + ruxolitinib
* Treatment B (N = 135): Capecitabine + placebo

Treatment consisted of repeating 21-day cycles. Capecitabine was self-administered for the first 14 days of each cycle, and ruxolitinib/placebo was self-administered during the entire cycle. Treatment for all participants was to continue as long as the regimen was tolerated, and the participant did not meet discontinuation criteria. Participants who discontinued treatment continued to be followed for subsequent anticancer treatments and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas.
* Advanced adenocarcinoma of the pancreas that is inoperable or metastatic.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Received 1 prior chemotherapy regimen for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy).
* ≥ 2 weeks elapsed from the completion of previous treatment regimen and participants must have recovered or be at a new stable baseline from any related toxicities.
* Radiographically measurable or evaluable disease
* An modified Glasgow Prognostic Score (mGPS) of 1 or 2 as defined below:

  * Criteria:

    1. mGPS of 1: C-reactive protein (CRP) > 10 mg/L and albumin ≥ 35 g/L
    2. mGPS of 2: CRP > 10 mg/L and albumin < 35 g/L

Exclusion Criteria:

* Received more than 1 prior regimen for advanced or metastatic disease.
* Ongoing radiation therapy, radiation therapy administered within 30 days of enrollment
* Concurrent anticancer therapy (eg, chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, hormonal therapy, investigational therapy, or tumor embolization).
* Current or previous other malignancy within 2 years of study entry without sponsor approval
* Prior severe reaction to fluoropyrimidines, known dihydropyrimidine dehydrogenase deficiency (DPD), or other known hypersensitivity to active substances, including fluorouracil (5-FU), ruxolitinib, or any of their excipients.
* Prior treatment with a JAK inhibitor for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, MD, Study Director — Incyte Corporation
Locations (95):
- United States (55):
  - Huntsville, Alabama
  - Fayetteville, Arkansas
  - Beverly Hills, California
  - La Jolla, California
  - Aurora, Colorado
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Macon, Georgia
  - Thomasville, Georgia
  - Harvey, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Minneapolis, Minnesota
  - Saint Louis Park, Minnesota
  - Bolivar, Missouri
  - Basking Ridge, New Jersey
  - Cherry Hill, New Jersey
  - Voorhees Township, New Jersey
  - Commack, New York
  - Fresh Meadows, New York
  - Harrison, New York
  - New York, New York
  - Rochester, New York
  - Rockville Centre, New York
  - Sleepy Hollow, New York
  - Canton, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Hershey, Pennsylvania
  - Langhorne, Pennsylvania
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Falls Church, Virginia
  - Newport News, Virginia
  - Seattle, Washington
  - Green Bay, Wisconsin
- Austria (5):
  - Graz
  - Linz
  - Salzburg
  - Vienna
  - Wein
- Chile (2):
  - Santiago
  - Vitacura
- Colombia (2):
  - Bogotá
  - Medellín
- Denmark (2):
  - Næstved
  - Odense C
- France (5):
  - Bordeaux
  - Brest
  - Dijon
  - Lyon
  - Nancy
- Ireland (3):
  - Cork
  - Dubin
  - Galway
- Israel (7):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
  - Tel Litwinsky
- Mexico (3):
  - Monterrey
  - Oaxaca City
  - Toluca
- Netherlands (3):
  - Amsterdam
  - Maastricht
  - Nijmegen
- Portugal (3):
  - Braga
  - Lisbon
  - Porto
- San Juan, Puerto Rico
- Sweden (2):
  - Linköping
  - Uppsala
- Switzerland (2):
  - Bellinzona
  - Geneva

REFERENCES:
- [Derived] Hurwitz H, Van Cutsem E, Bendell J, Hidalgo M, Li CP, Salvo MG, Macarulla T, Sahai V, Sama A, Greeno E, Yu KH, Verslype C, Dawkins F, Walker C, Clark J, O'Reilly EM. Ruxolitinib + capecitabine in advanced/metastatic pancreatic cancer after disease progression/intolerance to first-line therapy: JANUS 1 and 2 randomized phase III studies. Invest New Drugs. 2018 Aug;36(4):683-695. doi: 10.1007/s10637-018-0580-2. Epub 2018 Mar 6. PMID 29508247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced or metastatic adenocarcinoma of the pancreas who had failed or were intolerant to first-line chemotherapy were randomized in the study.
Pre-assignment Details: Treatment was started as soon as possible after randomization (within 3 days) and consisted of continuous 21-day cycles. Capecitabine was self-administered for the first 14 days of each cycle, and ruxolitinib/placebo was self-administered for the entire cycle.
Groups:
- Ruxolitinib Plus Capecitabine: Ruxolitinib 5 mg tablets in combination with Capecitabine 150 mg or 500 mg tablets to be administered by mouth twice daily (BID).
- Placebo Plus Capecitabine: Placebo 5 mg matching placebo tablets in combination with Capecitabine: 150 mg or 500 mg tablets to be administered by mouth twice daily (BID).
Period: Overall Study
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Started | 43 | 43
Completed | 3 (Treatment ongoing as of 13APR2016 for remaining participants in the study.) | 2 (Treatment ongoing as of 13APR2016 for remaining participants in the study.)
Not Completed | 40 | 41
Not completed — Disease progression | 26 | 27
Not completed — Adverse Event | 5 | 5
Not completed — Death | 3 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Other unspecified | 2 | 0
Not completed — Subject decision | 0 | 1
Not completed — Study Terminated by the Sponsor | 3 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.63) | 68.8 (8.43) | 67.1 (9.68)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 65 years | 20 | 13 | 33
  > 65 years | 23 | 30 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is reported here based on the number of deaths from randomization until the data cut-off.
Time Frame: Randomization until death due to any cause up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 43 | 43
Participants
  Observed deaths | 29 | 23
  Censored deaths | 14 | 20
Statistical Analysis 1: Comparison: Ruxolitinib Plus Capecitabine vs Placebo Plus Capecitabine; Test type: Other; Hazard Ratio (HR) = 1.584, 95% CI 2-sided [0.886 to 2.830]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause if sooner. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: Randomization to disease progression, or death due to any cause if sooner; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 43 | 43
days | 48.0 [37.0 to 83.0] | 61.0 [41.0 to 86.0]

3. Secondary Outcome: Percentage of Participants Achieving Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause if sooner. Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: as for outcome 2
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 43 | 43
percentage of participants
  Survival rate at 3 months | 0.337 [0.187 to 0.494] | 0.297 [0.157 to 0.451]
  Survival rate at 6 months | 0.131 [0.037 to 0.287] | 0.204 [0.088 to 0.352]

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate determined by radiographic disease assessments per Response Evaluation Criteria in Solid Tumours RECIST (v1.1), by investigator assessment and was defined as the percentage of participants with Complete Response (CR) or Partial Response (PR) by RECIST at any post baseline visit. Per RECIST for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline through end of study; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 43 | 43
percentage of participants
  Objective response | 4.7 | 2.3
  Complete response | 2.3 | 0.0
  Partial response | 2.3 | 2.3

5. Secondary Outcome: Duration of Response
Description: Duration of overall response was defined as the time in months from Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria in Solid Tumours (RECIST v1.1) until the first date Progressive Disease (PD) was objectively documented or until the date of death. Per RECIST for target lesions and assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target and non-target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions with no worsening of non-target lesions and no new lesions; Overall Response (OR) = CR + PR.
Time Frame: Baseline through end of study; up to 6-months or to the data cutoff 11FEB2016.
Population: The intent-to-treat (ITT) population consisted of all participants randomized to the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 43 | 43
days | NA [NA to NA] — The median duration of response was not evaluable in the treatment group due to the insufficient number of participants with events. | NA [NA to NA] — The median duration of response was not evaluable in the treatment group due to the insufficient number of participants with events.

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent AE was defined as an event occurring after exposure to at least 1 dose of study drug (ruxolitinib or placebo). A treatment-related AE was defined as an event with a definite, probable, or possible causality to study medication. A serious AE is an event resulting in death, hospitalization, persistent or significant disability/incapacity, or is life threatening, a congenital anomaly/birth defect or requires medical or surgical intervention to prevent 1 of the outcomes above. The intensity of an AE was graded according to the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 4.03: Grade 1 (Mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (life-threatening).
Time Frame: Baseline through approximately 30 days post treatment discontinuation; up to 6-months or to the data cutoff 11FEB2016.
Population: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug (ruxolitinib or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Number analyzed (Participants) | 42 | 43
Participants
  Participants who had any TEAEs | 41 | 40
  Participants who had treatment-related TEAEs | 21 | 25
  Participants who had SAEs | 28 | 20
  Participants who had Grade 3 or higher TEAEs | 31 | 31
  Participants hospitalized because of a TEAE | 26 | 18
  Participants discontinued treatment due to TEAE | 7 | 5
  Participants with a dose modification due to TEAE | 17 | 14
  Participants on concomitant medication due to TEAE | 36 | 35
  Participants with procedure performed due to TEAE | 22 | 14
  Participants who had a fatal TEAE | 8 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through the double-blind period through study termination up to 6-months or to the data cutoff 11FEB2016.
Description: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug (ruxolitinib or placebo).
Arm/Group | Ruxolitinib Plus Capecitabine | Placebo Plus Capecitabine
Serious Adverse Events (participants affected / at risk) | 28/42 | 20/43
Other Adverse Events (participants affected / at risk) | 38/42 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Plus Capecitabine (N=42) | Placebo Plus Capecitabine (N=43)
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Ascites (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Vascular disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 2
Sepsis (Infections and infestations) | 2 | 3
Cholangitis (Hepatobiliary disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Plus Capecitabine (N=42) | Placebo Plus Capecitabine (N=43)
Anaemia (Blood and lymphatic system disorders) | 16 | 10
Abdominal pain (Gastrointestinal disorders) | 14 | 4
Nausea (Gastrointestinal disorders) | 11 | 10
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12
Vomiting (Gastrointestinal disorders) | 10 | 10
Diarrhoea (Gastrointestinal disorders) | 10 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 10
Abdominal distension (Gastrointestinal disorders) | 10 | 4
Fatigue (General disorders) | 9 | 15
Constipation (Gastrointestinal disorders) | 8 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 10
Oedema peripheral (General disorders) | 7 | 8
Ascites (Gastrointestinal disorders) | 5 | 5
Pyrexia (General disorders) | 6 | 5
Asthenia (General disorders) | 7 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 3
Dizziness (Nervous system disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Blood bilirubin increased (Investigations) | 3 | 3
Anxiety (Psychiatric disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 6
Weight decreased (Investigations) | 3 | 4
Chills (General disorders) | 3 | 2
Oedema (General disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 3 | 0
Chest pain (General disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3
Hypotension (Vascular disorders) | 0 | 4
Blood creatinine increased (Investigations) | 0 | 3
Malaise (General disorders) | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain (General disorders) | 0 | 3
Platelet count decreased (Investigations) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
The study was terminated prior to the final analysis at the recommendation of the Data Monitoring Committee based on the review of efficacy in the 18424-362 (JANUS 1).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.